CLINICAL TRIAL: NCT01648530
Title: Chronic Migraine Epidemiology and Outcomes Study
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-BTX-12-470
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with Migraines: Participants who returned completed internet survey with positive screening for migraines. No intervention was administered in this study.
  Interventions: Other: No Treatment

INTERVENTIONS:
Other: No Treatment — No Treatment

SUMMARY:
This is a population internet-based study to characterize migraine clinical course and impact on family.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine
* U.S. Member of Survey Panel
* Household member of study participant
* Ability to complete internet-based questionnaires

Exclusion Criteria:

* No access to internet

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with migraine
Sampling Method: Non-Probability Sample
Enrollment: 16789 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan

REFERENCES:
- [Derived] Buse DC, Nahas SJ, Stewart WBF, Armand CE, Reed ML, Fanning KM, Manack Adams A, Lipton RB. Optimized Acute Treatment of Migraine Is Associated With Greater Productivity in People With Migraine: Results From the Chronic Migraine Epidemiology and Outcomes (CaMEO) Study. J Occup Environ Med. 2023 Apr 1;65(4):e261-e268. doi: 10.1097/JOM.0000000000002801. Epub 2023 Jan 25. PMID 36701797
- [Derived] Schwedt TJ, Buse DC, Argoff CE, Reed ML, Fanning KM, Hussar CR, Adams AM, Lipton RB. Medication Overuse and Headache Burden: Results From the CaMEO Study. Neurol Clin Pract. 2021 Jun;11(3):216-226. doi: 10.1212/CPJ.0000000000001037. PMID 34476122
- [Derived] Lipton RB, Fanning KM, Buse DC, Martin VT, Hohaia LB, Adams AM, Reed ML, Goadsby PJ. Migraine progression in subgroups of migraine based on comorbidities: Results of the CaMEO Study. Neurology. 2019 Dec 10;93(24):e2224-e2236. doi: 10.1212/WNL.0000000000008589. Epub 2019 Nov 5. PMID 31690685
- [Derived] Buse DC, Fanning KM, Reed ML, Murray S, Dumas PK, Adams AM, Lipton RB. Life With Migraine: Effects on Relationships, Career, and Finances From the Chronic Migraine Epidemiology and Outcomes (CaMEO) Study. Headache. 2019 Sep;59(8):1286-1299. doi: 10.1111/head.13613. Epub 2019 Aug 12. PMID 31407321
- [Derived] Adams AM, Serrano D, Buse DC, Reed ML, Marske V, Fanning KM, Lipton RB. The impact of chronic migraine: The Chronic Migraine Epidemiology and Outcomes (CaMEO) Study methods and baseline results. Cephalalgia. 2015 Jun;35(7):563-78. doi: 10.1177/0333102414552532. Epub 2014 Oct 10. PMID 25304766

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was an internet survey to identify participants with Episodic Migraine (EM) and Chronic Migraine (CM). The participants were followed for up to 1 year by assessments every 3 months.
Period: Overall Study
Arm/Group | Participants With Migraines
Started | 16789
Completed | 5915
Not Completed | 10874

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Migraines
Number analyzed (Participants) | 16789
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12495
  Male | 4294

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Episodic Migraine (EM) or Chronic Migraine (CM)
Description: EM is defined as <15 headache days/month and CM is defined as ≥15 headache days/month.
Time Frame: Baseline
Population: All qualified participants at Baseline who returned completed survey with positive screening for migraines.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Migraines
Number analyzed (Participants) | 16789
percentage of participants
  Episodic Migraine | 91.2
  Chronic Migraine | 8.8

2. Primary Outcome: Migraine Disability Assessment (MIDAS)
Description: The Midas score is a patient completed 5-item questionnaire about lost time and productivity (for work, school or family/social activities) in the past 3 months (number of days missed) where: 0-5=Little or No disability, 6-10=Mild disability, 11-20=Moderate disability or 21+ Severe disability. The Midas scores assessed at Months 3, 6, 9 and 12 were averaged.
Time Frame: 12 Months
Population: All qualified participants at Baseline who returned completed survey with positive screening for migraines.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Participants With Episodic Migraine: Participants who returned completed internet survey with Episodic Migraine defined as <15 headache days/month. No intervention was administered in this study.
- Participants With Chronic Migraine: Participants who returned completed internet survey with Chronic Migraine defined as ≥15 headache days/month. No intervention was administered in this study.
Arm/Group | Participants With Episodic Migraine | Participants With Chronic Migraine
Number analyzed (Participants) | 15313 | 1476
days | 13.1 (22.2) | 60.5 (70.4)

ADVERSE EVENTS:
Description: No Adverse Event data was collected in this study.
Arm/Group | Participants With Migraines
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No